CLINICAL TRIAL: NCT01572220
Title: Stress Echo Ultrasound Contrast in an Urban Safety Net Hospital to Refine Ischemia Evaluation
Acronym: SECURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Mori Krantz, Principal Investigator, Cardiologist, MD FACC FACP, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-0009
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Chest Pain; Symptomatic Ischemic Equivalent
Keywords: Hospitalized patients
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stress echocardiography (Other): Comparative effectiveness
  Interventions: Other: UCA stress echocardiography or myocardial SPECT
- Myocardial SPECT (Other): CER
  Interventions: Other: UCA stress echocardiography or myocardial SPECT

INTERVENTIONS:
Other: UCA stress echocardiography or myocardial SPECT — Comparative Effectiveness of cardiac stress imaging modalities

SUMMARY:
The current study is designed to have broad generalizability and inform a potential shift toward greater utilization of stress echocardiography with UCA. This will be accomplished by comparing UCA stress echocardiography with myocardial SPECT among hospitalized patients presenting with atraumatic chest pain. This study seeks to demonstrate: clinical comparability of the 2 modalities (based on non-diagnostic test rates), improved care efficiency (based on length of stay), lower costs, improved provider satisfaction, and a presumed improved safety profile through the elimination of radiation exposure.

Primary Hypothesis: A strategy of routine UCA (Optison™) enhanced stress echocardiography will result in a clinically non-diagnostic test rate comparable to myocardial SPECT among patients hospitalized (inpatient or hospital observation status) with atraumatic chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

  1. Males or females aged ≥ 18 years
  2. Evaluated for symptoms of chest discomfort or ischemic equivalent
  3. Clinical indication for stress imaging, defined as one of the following clinical risk estimates for CAD based upon the Diamond and Forrester classification7:

     * Intermediate pretest probability of CAD and electrocardiogram (ECG) is clinically interpretable and patient is able to exercise
     * Intermediate pretest probability of CAD and ECG is clinically interpretable or patient is unable to exercise
     * High pretest probability of CAD regardless of ECG interpretability and ability to exercise
  4. Willing and able to provide written informed consent to participate in this study
  5. Agrees to remain under observation (e.g., inpatient or observational status) until all study procedures from the hospital stay are completed, and to complete a 30-day follow up call

Exclusion Criteria:

* Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

  1. Documented medical history or discovery during screening and/or admission of any of the following:

     * Severe aortic or mitral stenosis
     * Significant resting left ventricular outflow tract obstruction (velocity > 3 cm/s)
     * Mobile left ventricular apical thrombus
     * Acute pericarditis or pericardial tamponade
     * Ascending or thoracic aortic aneurysm that is not stable or meets surgical criteria
     * Acute decompensated congestive heart failure
     * Established severe left ventricular systolic dysfunction (left ventricular ejection fraction < 35%)
  2. Definite acute coronary syndrome (e.g., unstable angina, acute myocardial infarction) as confirmed by elevated Troponin I (>0.6 ng/L) on two successive measurements or ECG changes diagnostic for unstable angina (e.g. localized ST changes) in conjunction with clinical appraisal
  3. Any of the following other abnormalities on the ECG at screening:

     * Paced ventricular rhythm or complete left bundle branch block
     * Uncontrolled arrhythmias defined by frequent premature ventricular complexes (PVCs) > 10/minute, non-sustained ventricular tachycardia, or atrial fibrillation with rapid ventricular response
     * 2nd or 3rd degree heart block
  4. Uncontrolled hypertension defined as systolic blood pressure ≥ 200 mmHg and/or diastolic blood pressure ≥ 110 mmHg at screening
  5. Hemoglobin (Hb) < 7.5 mg/dL at screening or within 3 months prior to screening
  6. Potassium < 3.0 mmol/L or > 5.5 mmol/L or severe electrolyte abnormality at screening that, in the opinion of the supervising physician or Investigator, makes stress testing unsafe
  7. Females who are pregnant or nursing
  8. Known intolerance to any of the study stress agents (dipyridamole, dobutamine) or study cardiac imaging agents (Optison, Cardiolite)
  9. Weight ≥ 350lbs
  10. Any physical or psychological condition that, in the opinion of the Investigator, may adversely affect the safety of the patient if enrolled in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Rate of non-diagnostic tests between ultrasound contrast enhanced stress echocardiography and myocardial SPECT | Within 5 days of stress imaging
  Non-diagnostic test rates will be the principal outcome of interest and are defined as those studies that do not allow a clinical decision for patient disposition (alternative non-invasive modality ordered, imaging inadequate to exclude ischemia, target heart rate not achieved, adverse side effects and test was terminated, discharge, further invasive testing such as coronary angiography) or require cardiology consultation for further evaluation.

SECONDARY OUTCOMES:
Similarity in rates of cardiac catheterization and acute coronary syndrome events between UCA stress echocardiography and myocardial SPECT | by 30 +/- 7 days post-discharge
  * 30-day rates of cardiac catheterization between the two imaging modalities
  * Difference in the 30-day composite rate of acute coronary syndrome re-hospitalization, revascularization, and death between the two imaging modalities
  * Similarity in positive predictive value (PPV) of the two imaging modalities
  * Inter-rater reliability estimates for non-diagnostic echocardiogram studies
Shorter length of stay and lower cost of inpatient hospital care for UCA stress echocardiography than for myocardial SPECT | 30 day assesment
  * Length of inpatient hospital stay of UCA stress echocardiography versus myocardial SPECT
  * Difference in time-to-cardiac catheterization beginning from time of admission
  * Differences in time-to-stress test completion beginning from time of admission30-day hospital costs of UCA stress echocardiography versus myocardial SPECT
Greater physician satisfaction when using UCA stress echocardiography than for myocardial SPECT | 5 days
  •Physician satisfaction as assessed on questionnaire with UCA stress echocardiography versus myocardial SPECT. Physician(s) will be the provider(s) who supervised patient care during inpatient hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Mori Krantz, MD FACC FACP, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Background] Garber AM, Solomon NA. Cost-effectiveness of alternative test strategies for the diagnosis of coronary artery disease. Ann Intern Med. 1999 May 4;130(9):719-28. doi: 10.7326/0003-4819-130-9-199905040-00003. PMID 10357690
- [Background] Berrington de Gonzalez A, Mahesh M, Kim KP, Bhargavan M, Lewis R, Mettler F, Land C. Projected cancer risks from computed tomographic scans performed in the United States in 2007. Arch Intern Med. 2009 Dec 14;169(22):2071-7. doi: 10.1001/archinternmed.2009.440. PMID 20008689
- [Background] Fazel R, Krumholz HM, Wang Y, Ross JS, Chen J, Ting HH, Shah ND, Nasir K, Einstein AJ, Nallamothu BK. Exposure to low-dose ionizing radiation from medical imaging procedures. N Engl J Med. 2009 Aug 27;361(9):849-57. doi: 10.1056/NEJMoa0901249. PMID 19710483
- [Background] Kisacik HL, Ozdemir K, Altinyay E, Oguzhan A, Kural T, Kir M, Kutuk E, Goksel S. Comparison of exercise stress testing with simultaneous dobutamine stress echocardiography and technetium-99m isonitrile single-photon emission computerized tomography for diagnosis of coronary artery disease. Eur Heart J. 1996 Jan;17(1):113-9. doi: 10.1093/oxfordjournals.eurheartj.a014669. PMID 8682117
- [Background] Diamond GA, Forrester JS. Analysis of probability as an aid in the clinical diagnosis of coronary-artery disease. N Engl J Med. 1979 Jun 14;300(24):1350-8. doi: 10.1056/NEJM197906143002402. PMID 440357
- [Derived] Salame G, Juselius WE, Burden M, Long CS, Bendelow T, Beaty B, Masoudi FA, Krantz MJ. Contrast-Enhanced Stress Echocardiography and Myocardial Perfusion Imaging in Patients Hospitalized With Chest Pain: A Randomized Study. Crit Pathw Cardiol. 2018 Jun;17(2):98-104. doi: 10.1097/HPC.0000000000000141. PMID 29768319
- See also: 6. ACCF/ASE/AHA/ASNC/HFSA/HRS/SCAI/SCCM/SCCT/SCMR 2011 Appropriate Use Criteria for Echocardiography — http://www.asecho.org/files/AUCEcho.pdf